CLINICAL TRIAL: NCT04584437
Title: The Treatment and Prevention of Covid-19 Infections Using Vitality Therapy or the Bible Cure
Brief Title: Treatment of Covid-19 Infections Using Vitality Therapy or the Bible Cure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Financial Support
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Principal Investigator, Dr. Kwasi Donyina, PhD, AMP, Founder and Chief Executive Officer, GAAD Medical Research Institute Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAADMRI
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Covid-19 Infections
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Prevention: The use of infrared sauna weekly will prevent COVID-19 infections. High doses of Vitamin C daily and supplements prevent Covid-19 infections. Drinking at least 4 litres of Vital Water daily will enhance ones health and prevent Covid-19 infections..
  Treatment: Infrared radiation for 60 minutes or the use of higher doses of Vitamin C as supplement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitality Therapy (Other): i. 500 to 1000 cubic centimeters of micro-clustered, hydrogen rich alkaline Vital Water.
  ii. Irradiation in infrared sauna for 60 minutes at high fever temperature. iii. Supplementation - Multivitamins and Minerals.
  Interventions: Other: Infrared Energy and Dietary Supplement

INTERVENTIONS:
Other: Infrared Energy and Dietary Supplement — Infrared Energy with a wavelength of 5 - 20 microns. Multivitamins and minerals including Vitamin C Supplements.

SUMMARY:
The human immune system is enhanced by exposure to infrared radiation with the wavelength of 5 microns to 20 microns. Humans, at normal body temperature, radiate most strongly in the infrared at a wavelength of about 10 microns. Infrared energy sustains life and can be used to treat and prevent diseases, including Covid-19 infections.

High temperature within the fever range obtained from infrared radiation causes the killer T-Cells to profilate. The Killer T-Cells improves ones immune system. The high temperature kills the Corona virus. In addition, multi-vitamins and minerals including high doses of Vitamin C, increase one's immune system. Vitamin C is an anti-oxidant, produces hydrogen peroxide and removes free radicals from the body.

Pre-clinical trials conducted in Houston, Texas, using Vitality Therapy or the Bible Cure were successful in curing Covid-19 infections.

It is therefore possible that Vitality Therapy or the Bible Cure can be used for the successful prevention and treatment of coronavirus infections.

DETAILED DESCRIPTION:
Dr. Donyina has successfully conducted 21 clinical trials and has discovered a three-pronged approach to prevention, treatment, and curing or management of all diseases. The medical protocols are based on:

1. Vital EnergyTM - Far Infrared with the wavelength of 5 to 20 microns,
2. Vital WaterTM - hydrogen-rich, micro-clustered, antioxidant, alkaline water is used to modify and enhance the pH of the human body, and;
3. Vital Minerals and Multi-VitaminsTM - proper nutrients enhance the healing process and prevent diseases.

   The three-pronged approach is known as Vitality TherapyTM or the Bible Cure for all curable and incurable diseases. God created a perfect body which can heal itself of any diseases thrown at it, provided the right environment exists. This environment is achieved by following the three-pronged approach to wellness and longevity. In addition, the 37.2 trillion mitochondria in the body are rejuvenated to provide energy and reverse the ageing process.

   Epigenetics documents that all medical conditions thought by the allopathic or conventional medical system to be due to genetics are now preventable and reversible by the three-pronged approach of Vital EnergyTM , Vital WaterTM, and Vital Minerals & Multi-VitaminsTM. In addition, the DNA script can perform at optimal levels to promote wellness.

   What is the difference between Drug Therapy (Pharmaceuticals) and Vitality TherapyTM or the Bible Cure (Drugless Therapy) approach to disease control, prevention, and treatment?

   The paradigm characterizing drug therapy (i.e., using pharmaceuticals) is as follows: for a specific disease, drugs or radiations are used for treatment. Thus, the treatments are disease specific. So, if one has cancer, one may use Chemotherapy for cancer treatment. If one has another disease such as diabetes, Chemotherapy will be of no use. One must use a drug that is specific for diabetes, such as insulin or an oral agent like Metformin HCl (Glucophage®).

   There is a new drugless paradigm, which can be exemplified by strengthening the human immune system. The human body is capable of healing itself from any disease thrown at it provided the immune system is heightened. Our focus is to strengthen the immune system by providing the body the energy and essential plant-based and sea food nutrients it requires for repairs and growth in an optimum pH environment. The external energy is provided by vital energyTM medical devices and the optimum pH environment is achieved by drinking vital waterTM produced by medical devices. The nutrients are mainly plant and seafood based enriched with multi-vitamins and minerals. Acidic foods, like beef, are generally avoided.

   Thus, the paradigm shift is from disease-specific treatment offered by allopathic medical practitioners and Big Pharma to enhancing the human immune system for the treatment of curable and incurable diseases. We strongly believe that all diseases are curable because of the heightened immunity. Let us compare Drug Therapy with Drugless Therapy:

   DRUG THERAPY (Odd #s) VITALITY THERAPY or the Bible Cure (Even #s)

   (1). Based on artificial chemicals (2). Plants, vitamins, minerals, micro clustered antioxidant and hydrogen-rich alkaline water, and infrared energy

   (3). Artificial therapy (4). Natural therapy

   (5). Generally, destroys human life (6).Sustains human life

   (7). Destroys human immunity (8).Enhances human immunity

   (9). Acidifies the human body (10). Alkalizes the human body

   (11). Induces diseases (e.g., Dexamethasone Induces Diabetes) (12). Heals curable and incurable diseases

   (13). Causes the ageing of the body (14). Reverses ageing

   (15).. Oxidizes the body (16).Anti-oxidation of the human body

   (17). Toxic chemicals (18).Natural products

   (19). Destroys brain and nerve cells (20). Brain and nerve cells are regenerated

   (21). Destroys cartilage, causing arthritis (22).Regrows cartilage, thus cures arthritis

   (23). Feeds cancerous cells (24).Destroys cancerous cells

   (25). Causes neurodegenerative diseases (26).Cures neurodegenerative diseases

   (27). Causes neuromuscular disorders (28).Cures neuromuscular disorders

   (29). Destroys mitochondria in the body (20).37.2 trillion mitochondria are rejuvenated to provide energy and reverse the ageing process

   (31). Numerous side effects. The drugs and the side effects will, in general, cause death (32). NO SIDE EFFETS

   (33). Approximately 80% of allopathic medicine is quackery. (34)Actual curing of diseases and no quackery

   Let us briefly examine quackery in allopathic medicine. An othopedic surgeon performs knee sugery at the cost of over $10,000 dollars. Vitality Therapy or the Bible Cure treats arthritis with Shark Cartilage. The cost is less that $200. The cartilage grows back. In addition, far infrared energy regrows worn out cartilage.

   Cancer

   Chemotherapy is generally used to treat cancer. It is noteworthy that chemotherapy is very strong toxic chemical and kills both good and cancerous cells. The survival rate is less than 10% at an exorbitant cost to insurance companies and governments. Allopathic practitioners and Big Pharma earn trillions of dollars annually while KILLING PATIENTS because drug therapies do not cure diseses.

   Vitality Therapy or the Bible Cure treats all stages of cancer with no side effects. The body is changed from being acidic to basic. Thus the cancer cells, which cannot survive in the basic environment, and are killed. The high temperature environment provded by infrared energy also kills cancerous cells. Treatment cost for cancer is minimal.

   Drugs do not cure diseases but just minimize the symptoms. Vitality TherapyTM or the Bible Cure enhances the immune system for the healing of all diseases and also provides longevity and disease-free living.

   SCIENTIFIC EXPLANATION - VIROLOGY & IMMUNOTHERAPY
   1. Hirayama E. et al. J. Virology 2004 (Virology)

      This paper is the key to how sauna therapy works against RNA viruses, including Covid-19. Heat shock protein-70 (HSP70) is increased by sauna therapy and inhibits viral protein export and replication.

      Thus heat kills Covid-19. Please note that there is no Covid-19 in Desert Areas or Tropical Countries. Covid-19 is imported from cold climate countries to desert and tropical countries.
   2. IMMUNOTHERAPY (High Temperature and Multivitamins and Minerals + Vitamin C)

   The immune system is enhanced by infrared energy which increases the body temperature. The normal body temperature is approximately 36.5 - 37.5 degrees C. Vital energy irradiation increases the body temperature to the range of 37.5 - 39 degrees C which is equivalent to fever temperature. The temperature could even be higher than 39 degrees C or high fever range, depending on the temperature setting of the infrared sauna. The high body temperature causes an unbearable environment for some pathogens and viruses. Killer T-cells also rapidly proliferate due to the suitable environment and can also help fight off the harmful viruses, pathogens and microbes that have invaded the body.

   The body temperature in the fever range has several important functions in the healing process including, but are not limited to the following:

i. increased mobility of leukocytes ii. enhanced leukocytes phagocytosis iii. endotoxin effects decreased iv. increased proliferation of T Cells v. enhanced activity of interferon

Multivitamins and Minerals (+Vitamin C)

High doses of Vitamin C kills pathogens, viruses and disease-causing microbes. High doses of Vitamin C increases one's immune system. Vitamin C is an anti-oxidant, produces hydrogen peroxide and removes free radicals from the body. Vitamin C has several other medical benefits including repairing damaged tissues and organs.

During the cold season, one should use high doses of Vitamin C (5 gm to 10 gm, depending on the body weight, daily) to prevent and treat colds and influenza.

The only side effect of high doses of Vitamin C that I am aware of is that it may cause diarrhea. However, diarrhea is a good way to clean and detoxify the body.

Some experts interpret the prevalence of Covid-19 pandemic worldwide based on:

1. Youthful demographics
2. Altitude
3. Warmer temperatures
4. Poorer communities

   Condition (3) above (i.e. Temperature) was dismissed. It is my opinion that warmer temperatures play critical role in the control, management and treatment of the coronavirus.

   i. Asia, Europe and North America have pronounced peaks because of cold temperature. A second wave of the pandemic is hence, expected in winter months.

   ii. It is believed that, Latin America and the Caribbean have peaks as a result of poorer communities (over crowding).

   iii. Middle East and Africa have low cases because of warmer temperatures. This is supported by the temperature effects on coronavirus (Virology) and heightened immune system when the human body is subject to high temperature (immunotherapy).

   SUMMARY OF VITALITY THERAPY OR THE BIBLE CURE FOR ALL DISEASES

   The fundamental principles underlying the Bible Cure or the three-pronged approach to wellness, longevity and disease-free living are as follows:

   i. Humans are living energies and the energy level must be kept as high as possible; ii. What we eat is ultimately what determines our health, energy level and the state of our body and alkaline diet is essential to our wellness; iii. The human body shall be kept in an alkaline condition (pH of 7.3 to 7.4) as pathogens and viruses generally cannot exist in alkaline medium (Blood pH is 7.365); iv. Water is critical to good health. Humans are approximately 75% water. Water purity, its alkalinity and anti-oxidative properties are important to health; v. Multi-Vitamins and minerals are essential to our wellness; vi. We cannot eliminate stress from our lives. However, we can learn how to manage it; and, vii. Exercise must be part of our daily routines.

   It must be noted that these toxic pharmaceuticals do not CURE diseases.

   Given the right environment, the body can cure itself of whatever disease thrown at it, hence disease-free living and longevity are achieved.
   * The effects of ageing are reversed, and the oxidation of the human cells are prevented, thus one becomes young again;
   * The therapy provides the much-needed energy to the nervous system and the whole body;
   * Improves the autonomic functions of the nervous system;
   * Improves and restores the functions of the endocrine system;
   * Restores the body's communication system;
   * Strengthens the immune system;
   * Improves of blood circulation;
   * Increases the level of oxygen in the cells;
   * Promotes the regeneration of cells and fast healing;
   * Activates the water molecules in the body;
   * Brain and nerve cells are regenerated;
   * Pain management - analgesic effect of vital energy;
   * Destroys cancerous (e.g. breast cancer) and benign (e.g. uterine fibrous) tumors;
   * Autoimmune diseases like diabetes and HIV/Aids have responded well to Vitality Therapy™ or the Bible Cure
   * Neurodegenerative diseases respond positively to the Vitality Therapy™ (Alzheimer's disease and Multiple Sclerosis);
   * There are beneficial effects on neuromuscular disorders (i.e. muscular dystrophies),
   * Vitality Therapy™ or the Bible Cure has no side effects as vital energy sustains life and is the same energy obtained from food during respiration, and;
   * The 37.2 trillion mitochondria in the body are rejuvenated to provide energy and reverse the ageing process.

   CONCLUSION

   We strongly believe that Vitality Therapy or the Bible Cure can prevent and cure Covid-19 infections. Our pre-clinical trials in Houston, Texas, USA were very successful. Patients were completely cured.

ELIGIBILITY:
Inclusion Criteria:

* All humans seeking prevention or treatment of the COVID-19 pandemic.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-25 (Estimated); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-07-10 (Estimated)

PRIMARY OUTCOMES:
Treatment and Prevention of COVID-19 Pandemic. | 10 months
  The Use of Infrared Energy and Vitamin C Supplement for the Treatment and Prevention of COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- GAAD Medical Research Institute Inc. O/A The Centre for Incurable Diseases, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No